CLINICAL TRIAL: NCT05787197
Title: Circulating Tumor DNA in Patients With Colorectal Cancer Undergoing Curative-intent Surgery for Liver Metastases: Prospective, Multicenter, GERCOR Cohort
Brief Title: ctDNA in CRC Patients Undergoing Curative-intent Surgery for Liver Metastases
Acronym: CLIMES
Status: Recruiting | Type: Observational
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Other Study IDs: CLIMES G-118 CIRCULATE-4
Record Dates: First submitted 2023-03-08; First posted 2023-03-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer; Circulating Tumor DNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected in the pre-operative setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective multicenter cohort study, was designed to explore the prognostic value of ctDNA as a biomarker of disease response and recurrence or death in patients undergoing curative-intent surgical resection of Colorectal cancer liver metastasis.

DETAILED DESCRIPTION:
Blood collection times according to specific clinical situations:

* Standard approach
* Combined surgery
* Reverse strategy
* Two-stage hepatectomy

ELIGIBILITY:
Inclusion criteria

The patient will be included if:

1. Has signed informed consent form and is willing to comply with all study procedures and availability for the study duration,
2. Is ≥ 18 years of age,
3. Has histologically confirmed colorectal adenocarcinoma,
4. Has resected primary tumor or is eligible to primary tumor and CRLM (in case of synchronous metastases) resection within 6 months prior to study inclusion,
5. Has isolated CRLM that is deemed resectable or potentially resectable (extrahepatic metastases excluded, except infracentimetric non-specific lung lesions with largest diameter <1 cm and maximal number of ≤3) as judged by a multidisciplinary team meeting (based on CT scans of chest, abdomen, and pelvis [or MRI if CT not possible]),
6. Is eligible to surgical procedure,
7. Is fit for the chemotherapy-surgery combination treatment,
8. Is registered in a national health care system (Protection Universelle Maladie [PUMa] included).

Exclusion criteria

The patient will be excluded if:

1. Has definitively unresectable CLRM,
2. Had more than 9 pre-operative cycles of chemotherapy for treatment of metastatic disease planned at inclusion,
3. Has not resected primary rectal tumor (low and middle),
4. Has history of another primary cancer within the last 5 years, with the exception of non-melanomatous skin cancer and carcinoma in situ of the cervix,
5. Has no more than two surgical procedures planned for complete resection of primary tumor and/or liver metastases,
6. Has deficient mismatch repair (dMMR)/ microsatellite instability (MSI) tumors treated with immunotherapy,
7. Blood samples cannot be collected if surgical procedure,
8. Is pregnant or breastfeeding,
9. Cannot be followed-up due to geographical, social, or psychic conditions,
10. Has medical or psychiatric condition or occupational responsibilities that may preclude compliance with the protocol,
11. Is under guardianship, curatorship, or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active file in oncology department
Sampling Method: Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) in patients who undergo curative-intent resection of colorectal liver metastasis (CRLM) | Up to 36 months
  DFS is defined as the time from complete surgical resection (following first surgery if one-stage surgery or second surgery if two-stage strategy) to first documented event (relapse or death, whichever occurred first), or until last contact if no event occurs.

SECONDARY OUTCOMES:
Number of event-free survival (EFS) in patients who undergo curative-intent resection of CRLM. | Up to 4 years
  EFS is defined as time between inclusion until the occurrence of an event: disease progression, relapse, disease progression, or death from any reason.
Overall survival (OS) n patients who undergo curative-intent resection of CRLM. | Up to 4 years
  OS is defined as the time between inclusion and death. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period.
Time to surgical failure (TSF) in patients who undergo curative-intent resection of CRLM. | Up to 4 years
  TFS is defined as the time from initial surgery until the first unresectable recurrence or death from any cause or the date of the last follow-up, at which point data are censored.
Prognostic value of ctDNA | Up to 4 years
  Prognostic value of ctDNA:
  * post-operative ctDNA detection,
  * relative change in ctDNA level after curative resection of CRLM,
  * ctDNA in different subgroups of patients classified according to the type of surgical strategy (standard approach, combined surgery, reverse strategy, two-staged hepatectomy),
Prognostic factor(s) for disease recurrence and survival. | Up to 4 years
  Prognostic factor(s) for disease recurrence and survival in patients who undergo curative-intent resection of CRLM.
Association between ctDNA and clinical features. | Up to 4 years
  To identify the clinical, biological, and pathological factors associated with the ctDNA level.

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano GELLI, MD, Principal Investigator — Department of Digestive Surgery, Gustave Roussy Hospital
Locations (16):
- France (16):
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Lille - Hôpital Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Bichât Claude Bernard, Paris
  - Hôpital Cochin, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Haut Lévêque, Pessac
  - CHU de Poitiers, Poitiers
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHRU Tours, Tours
  - Hôpital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif